CLINICAL TRIAL: NCT03178383
Title: Integration of Cancer Health Activities Into African American Churches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: American Cancer Society, Inc. (Other); Community Ministry of Prince George's County (Unknown); Access to Wholistic and Productive Living Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RSG-16-022-01-CPPB
Record Dates: First submitted 2017-05-18; First posted 2017-06-06 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer; Prostate Cancer; Colorectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Approach (Experimental): In this approach, rather than developing a separate health ministry, cancer activities could be integrated throughout existing church ministries (e.g. men's, women's, seniors).
  Interventions: Behavioral: Project HEAL 2.0
- Standard Comparison (Active Comparator): Standard group churches will not be asked to, or provided special encouragement to technical assistance with, institutionalizing health promotion activities in their churches.
  Interventions: Behavioral: Project HEAL

INTERVENTIONS:
Behavioral: Project HEAL — Standard group churches will not be asked to, or provided special encouragement to technical assistance with, institutionalizing health promotion activities in their churches.
  Arms: Standard Comparison
Behavioral: Project HEAL 2.0 — In this approach, rather than developing a separate health ministry, cancer activities could be integrated throughout existing church ministries (e.g. men's, women's, seniors).
  Arms: Integrated Approach

SUMMARY:
The proposed project will compare two ways to apply a known-effective cancer educational strategy through African American churches: 1) a standard method vs. 2) a new method in which the churches integrate the strategy into their organizational structure and practice at multiple levels. It will be determined whether this "integrated approach" results in more effective and sustained cancer education and screening activities at both the church and individual levels over time. This project will make important contributions to research in evidence-based medicine and sustainability. In a climate of limited resources, identifying sustainable and effective ways to increase cancer awareness and screening in African American men and women is more important than ever.

DETAILED DESCRIPTION:
This population-based application responds to the American Cancer Society Research Scholar Grant, Priority Program in Cancer Control. Recent years have seen a growing research interest in learning how to get known-effective health education strategies to reach more people who could benefit from them. An important part of this growing movement is a focus on sustained impact, or continued program benefit after the funding period is over. It is believed that the best way to achieve this sustained impact is through integrating the program into the host community at multiple levels. This innovative strategy has not been systematically tested in community-based settings, where the most vulnerable people can be reached. Since churches have a historical and ever-growing role in health promotion particularly among African Americans, they are an ideal place to reach this group for cancer education. The proposed project will compare two ways to apply a known-effective cancer educational strategy through African American churches: 1) a standard method vs. 2) a new method in which the churches integrate the strategy into their organizational structure and practice at multiple levels. It will be determined whether this "integrated approach" results in more effective and sustained cancer education and screening activities at both the church and individual levels over time. The educational strategy is one that has been used successfully in previous work: Project Health through Early Awareness and Learning (HEAL). Project HEAL is a series of three cancer early detection workshops (breast, prostate, colorectal) delivered through trained and certified lay peer community health advisors in African American churches. 14 churches will be randomly chosen to conduct either the standard Project HEAL program or an integrated Project HEAL strategy where the churches build the program into their organization in multiple ways (e.g., allocating volunteer or paid staff, space, or funds; policy change; ministry development). The project will be conducted in three phases: 1) refining the integrated approach with community and stakeholder feedback; 2) pilot testing the integrated approach in 2 churches; and 3) conducting the study to comparatively evaluate the standard vs. the integrated approaches in 14 churches. A scientifically rigorous evaluation plan will be used to look at outcomes at both the individual and the church level. This project will make important contributions to research in evidence-based medicine and sustainability. In a climate of limited resources, identifying sustainable and effective ways to increase cancer awareness and screening in African American men and women is more important than ever.

ELIGIBILITY:
Inclusion Criteria:

* Advisory Panel members: adults ages 21+
* Pastors, representing each of the 14 churches enrolled in the project: active pastor of churches enrolled in the study
* Community Health Advisors
* Self-identified African American
* Adults ages 21+
* Regularly attend church services
* Able to complete Project HEAL training
* Able to recruit 40+ participants for a breast, prostate, or colorectal cancer educational workshop
* Able to lead the breast, prostate, and colorectal cancer workshops
* Workshop Participants
* Self-identified African American
* Adults ages 21+
* Have no history of breast, prostate, or colorectal cancer

Exclusion Criteria:

* Workshop Participants: Men and women who have had breast, prostate, or colorectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Integration of health-relation practices assessed via church survey | Change from baseline to 12 and 24 months
  Intervention impact on institutionalization at 12 and 24 months

SECONDARY OUTCOMES:
Reach: Number of participants from priority population engaged in intervention as assessed by enrollment logs | Up to 4 months
  Participants from priority population engaged in intervention
Efficacy: Increased knowledge of cancer as assessment by participant surveys | Up to 12 months
  Cancer-related knowledge
Efficacy: Increased self-report of cancer screening as assessment by participant surveys | Up to 12 months
  Self-reported cancer screening
Adoption | At recruitment/enrollment
  Cooperation rate of churches
Implementation: Extent to which intervention is implemented as intended as assessed by a fidelity checklist completed by staff | Up to 4 months
  Adherence to intervention protocol

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl L Holt, PhD, Principal Investigator — Professor
Locations (1):
- University of Maryland School of Public Health, College Park, Maryland, United States

REFERENCES:
- [Derived] Knott CL, Chen C, Bowie JV, Mullins CD, Slade JL, Woodard N, Robinson-Shaneman BR, Okwara L, Huq MR, Williams R, He X. Cluster-randomized trial comparing organizationally tailored versus standard approach for integrating an evidence-based cancer control intervention into African American churches. Transl Behav Med. 2022 May 26;12(5):673-682. doi: 10.1093/tbm/ibab088. PMID 34255087
- [Derived] Knott CL, Bowie J, Mullins CD, Santos SLZ, Slade J, Rosenberg E, Woodard N, Williams R, Williams RM. An Approach to Adapting a Community-Based Cancer Control Intervention to Organizational Context. Health Promot Pract. 2020 Mar;21(2):168-171. doi: 10.1177/1524839919898209. Epub 2020 Jan 20. PMID 31959002
- See also: CHAMP Lab Website — http://bit.ly/CHAMPLab